CLINICAL TRIAL: NCT00289549
Title: Phase II Study of Forodesine Hydrochloride in Patients With Advanced, Fludarabine-Refractory Chronic Lymphocytic Leukemia (CLL)
Brief Title: Study of Forodesine Hydrochloride in Patients With Advanced, Fludarabine-refractory Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCX1777-Bo-05-204
Record Dates: First submitted 2006-02-08; First posted 2006-02-10 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Leukemia, Lymphocytic, Chronic
Keywords: CLL; Chronic lymphocytic leukemia; leukemia; Advanced, fludarabine-refractory CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia | interventions — forodesine

INTERVENTIONS:
Drug: forodesine hydrochloride (BCX-1777) — experimental, forodesine oral dose 200 mg administered daily.

SUMMARY:
Forodesine hydrochloride will be administered orally at a dose of 200 mg daily for 7 days each week for 4 weeks (cycle number 1). The drug will be administered once daily one hour prior to or two hours after meals. Patients will be evaluated after 1 full cycle of therapy (28 days).

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 years and older
* Diagnosis of CLL established by peripheral blood and bone marrow examination and using the standard criteria
* Patients with Rai stage III or IV, or earlier stage with massive, symptomatic lymphadenopathy requiring therapy
* Primary resistance to fludarabine-based therapy (no complete response [CR] or partial response [PR]) or progressive disease within 6 months of response to prior fludarabine containing regimen.
* ECOG performance status of 0, 1, 2 or 3
* Willing to take adequate contraception (i.e. latex condom, cervical cap, diaphragm, abstinence, etc.) for the entire duration of the study and 3 months after
* All investigational treatments should have been discontinued for at least 1 week prior to the initiation of the study drug.

Exclusion Criteria:

* Pregnant or nursing
* Unable or unwilling to sign consent
* Severe, ongoing co-morbid conditions, which would preclude safe delivery of the investigational therapy
* Active serious infections that are not controlled by antibiotics
* ECOG performance status 4
* Inadequate renal function: creatinine 2.0 or more unless related to the disease
* Inadequate liver function: bilirubin 3.0 or more, transaminases 3 x upper limit of normal or more unless related to the disease
* Known positive test for HIV
* Patients with known hepatitis B and/or hepatitis C active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2005-06; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Response rate after 2 cyclesof forodesine therapy. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Ravandi, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, University of Texas, Houston, Texas, United States

REFERENCES:
- [Derived] Balakrishnan K, Verma D, O'Brien S, Kilpatrick JM, Chen Y, Tyler BF, Bickel S, Bantia S, Keating MJ, Kantarjian H, Gandhi V, Ravandi F. Phase 2 and pharmacodynamic study of oral forodesine in patients with advanced, fludarabine-treated chronic lymphocytic leukemia. Blood. 2010 Aug 12;116(6):886-92. doi: 10.1182/blood-2010-02-272039. Epub 2010 Apr 28. PMID 20427701